CLINICAL TRIAL: NCT05143801
Title: "Facemask Use During High-intensity Interval Exercise in Temperate and Hot Environments"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Christine Mermier PhD, Professor, University of New Mexico
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 1680206
Record Dates: First submitted 2021-10-24; First posted 2021-12-03 (Actual); Results first posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-03

CONDITIONS: Hypoxemia; Physiological Stress
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Intervention Model Description: non-blinded randomized repeated measures crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- No mask temperate (Active Comparator): Participant exercised in room temperature environment not wearing a surgical face mask
  Interventions: Other: High-intensity interval exercise without using a surgical face mask in a temperate environment
- Mask temperate (Experimental): Participant exercised in room temperature environment while wearing a surgical face mask
  Interventions: Device: High-intensity interval exercise with surgical face mask in a temperate environment
- No mask hot (Active Comparator): Participant exercised in a hot environmental temperature not wearing a surgical face mask
  Interventions: Other: High-intensity interval exercise without using a surgical face mask in a hot environment
- Mask hot (Experimental): Participant exercised in a hot environmental temperature while wearing a surgical face mask
  Interventions: Device: High-intensity interval exercise with surgical face mask in a hot environment

INTERVENTIONS:
Device: High-intensity interval exercise with surgical face mask in a temperate environment — Participants performed high-intensity interval exercise in a temperate environmental condition while wearing surgical face mask
  Arms: Mask temperate
Device: High-intensity interval exercise with surgical face mask in a hot environment — Participants performed high-intensity interval exercise in a hot environmental condition while wearing surgical face mask
  Arms: Mask hot
Other: High-intensity interval exercise without using a surgical face mask in a hot environment — Participants performed high-intensity interval exercise in a hot environmental condition without wearing a surgical face mask
  Arms: No mask hot
Other: High-intensity interval exercise without using a surgical face mask in a temperate environment — Participants performed high-intensity interval exercise in a temperate environmental condition without wearing a surgical face mask
  Arms: No mask temperate

SUMMARY:
To investigate surgical mask use and high-intensity interval exercise across different environmental conditions.

DETAILED DESCRIPTION:
Mask use in public settings is recommended to limit the spread of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) that causes the disease known as COVID-19 and endorsed by the Centers for Disease Control and Prevention (CDC) and the World Health Organization (WHO). Wearing a mask during exercise may have implications for recreational exercisers and athletes that train and compete at a high exercise intensities as it has been shown to limit ventilation (VE) and increase end-tidal CO2 compared to a no-mask control. For example, N95 masks are designed to fit more tightly around the nose and mouth than other types of masks and have been shown to reduce markers of maximal exercise performance compared to a no-mask control for individuals performing an incremental ramp protocol on a cycle ergometer.

In contrast to N95 masks being reserved for health care workers, surgical masks certified by National Institute for Occupational Safety and Health are easily accessible to wear during exercise to reduce the risk of COVID-19 spread. Indeed, these masks fit more loosely than the N95, but did not reduce maximal power (Pmax), relative oxygen consumption (mL/kg/min), or test duration in two studies where participants performed a progressive maximal exercise test on a cycle ergometer. Further, surgical mask use during a progressive maximal cycling exercise protocol did not change cardiovascular, metabolic, and pulmonary measurements when compared to a no-mask condition in healthy individuals, with the exception of a decrease in maximal heart rate (HRmax). Another recent study using a progressive maximal cycling exercise protocol showed no change in (HRmax) using cycle ergometry when surgical mask use was compared to a no-mask condition. While this type of progressive maximal exercise test is frequently used for clinical and laboratory settings to assess cardiovascular, pulmonary, and metabolic markers, this type of exercise protocol is not often employed by athletes seeking to improve performance or recreational exercisers taking action to improve fitness. Because this exercise protocol is not used by athletes or recreational exercisers to train, it is difficult to translate the results of mask use during progressive maximal exercise tests to commonly practiced forms of exercise. In fact, a recent meta-analysis concludes that wearing a mask elicits a minimal impact on cardiovascular, respiratory, or metabolic variables across a wide array of exercise intensities and modalities, however, high intensity interval exercise (HIIE) was not included in this analysis, nor were hot environmental temperatures. Thus, the physiologic or metabolic responses while wearing a medical-grade surgical mask are not yet known with HIIE in both temperate and hot environments.

High intensity interval exercise is a popular time-efficient training method that involves short high intensity bouts followed by either active (low/moderate intensity exercise) or passive (no exercise) rest bouts. High intensity interval exercise has been shown to be a safe and effective way to increase physical fitness or performance in a diverse population that include exercisers in recreational, competitive, and clinical settings. Further, as HIIE can be performed in either an indoor or outdoor environment and using a mask may increase the physiological and perceptual strain of the exercise depending on the temperature and humidity. In a hot environment (40°C and 20% humidity), no difference was found in skin temperature under or outside a KN95 mask in healthy males that performed 45-minutes of moderate intensity physical activity that mimicked movements required in occupational settings. Also, no difference was found in whole body thermal discomfort, and an increase in perceived breathlessness by 36% was observed. In addition, surgical mask use during 30 minutes of mild uphill treadmill exercise did not increase risk of heat stroke in a hot and humid environment. To date, no research study has investigated the effects of surgical mask use during HIIE in different environmental conditions.

Therefore, the purpose of this study was to investigate the effects of surgical mask use during HIIE on cardiovascular, metabolic, thermoregulatory, and perceptual responses in temperate and hot environments.

Methodsː In a randomized fashion, ten healthy participants completed two HIIE sessions in a 36°C hot (HIIE-HOT) and two HIIE sessions in a 23°C temperate environment (HIIE-TEMP) while wearing (MASK) and not wearing a surgical mask (CON).

Procedures Anthropometrics and maximal Oxygen uptake measurements Before the experimental trials, participants visited the Exercise Physiology laboratories for anthropometrics and VO2max measurement. Body height was measured using a stadiometer (SECA, seca 216, Chino, CA, USA) and weight was measured using a digital scale (Cardinal DETECTO 758C, Webb City, MO). Then, participants completed a 5-minute warm-up at a self-selected exercise intensity prior to the VO2max test on an electrically braked cycle ergometer (Lode, Excalibur Sport, Groningen, The Netherlands). During the VO2max test, HR was measured using a Polar HR monitor (Polar, Polar H10, USA) with each test designed to last between 10 and 12 minutes. The starting resistance and the continuous increase in resistance (between 20-40 watts) throughout the test was based on the participants' self-reported fitness. Termination of the VO2max test occurred at volitional fatigue or when the participant could no longer maintain a cycling cadence of 60 revolutions per minute or higher. Gas-exchange was measured using a metabolic analyzer (Parvo Medics Inc, TrueOne 2400, Salt Lake City, UT) and data were analyzed using an 11-breath rolling average20. Primary criteria for a VO2max was categorized as an observed plateau that varied by less than 150 mlO2/min21. To determine a plateau using primary criteria, the mean of the absolute difference from each neighboring data point in the last 30 seconds of the 11-breath rolling average VO2 was compared against 150 mlO2/min21; if the average value was smaller, the test was categorized as a VO2max. In the absence of a plateau, a VO2max was confirmed if two of the three secondary criteria were met: 1) an RPE ≥17, 2) a respiratory exchange ratio (RER) of 1.1 or greater, and 3) a HR within 10 beats of estimated heart rate max using the Jones et al. equation (202 - 0.72 x age). The highest power output recorded from the VO2max test was used to calculate the high intensity and active recovery bouts for the HIIE sessions.

High Intensity Interval Exercise Trials Before all HIIE sessions participant's hydration status was assessed measuring urine specific gravity (USG) using a handheld refractometer (Cole-Parmer, RSA-BR90A, Vernon Hills, IL). A USG measurement lower than 1.020 g/cc allowed participants to proceed to the HIIE sessions. If USG was greater than 1.020 g/cc, then participants consumed 500 ml of water, and were reassessed after 30 minutes. This water provision was only repeated twice if USG remained above 1.020 g/cc.

A randomized cross over repeated measures design was used to compare cardiovascular, thermoregulatory, metabolic, and perceived responses before and during HIIE across four experimental trials performed during two visits. For each visit, which was separated by a minimum of 72 hours, the participants completed two HIIE sessions separated by 3 hours of rest. Each HIIE bout consisted of 10 bouts lasting 30 seconds performed at 85% Pmax followed by 90 seconds of active recovery at 30% Pmax. The HIIE sessions were performed in a temperate environment (23°C, 25% relative humidity) with (TEMP/MASK) and without a surgical mask (TEMP/CON), and in a hot environment (36°C, 14% relative humidity) with (HOT/MASK) and without a surgical mask (HOT/CON). During the exercise protocol participants were allowed to drink water.

During HIIE sessions with a mask, all participants were instructed to wear the surgical mask snugly over their nose and mouth. The participants fitted the flexible metal plate within the surgical mask over the bridge of the nose and had the bottom of the mask cover underneath the chin. During the 3-hour rest period participants were provided a 350-calorie meal (7g of Fat; 64g Carbohydrate; 9g Protein) and water ad libitum.

Cardiovascular Measurements Before every HIIE trial and after 5-minutes of seated rest, resting blood pressure was measured using a sphygmomanometer, and stethoscope. A cardiac impedance device (PhysioFlow®, NeuMeDex, Bristol, PA) calibrated per manufacturer guidelines was used to indirectly measure cardiac output (CO), stroke volume (SV), and HR. These measurements were taken continuously using 10-second averaging provided by the PhysioFlow® software during each HIIE session.

Metabolic Measurements A near infra-red spectroscopy (NIRS) device (Moxy, Moxy Monitor System, MN, USA) was used to measure muscle tissue oxygenation every second during each HIIE session. The highest muscle tissue oxygenation value from each active rest period (MTO active rest %) was averaged for each HIIE session. Additionally, the lowest muscle tissue oxygenation (MTO during HIIE %) value per high intensity bout was recorded and averaged from each HIIE session. The difference of the average MTO active rest % and MTO during HIIE % was used to calculate the muscle tissue oxygenation difference (MTO difference %). All MTO measurements were taken on the dominant leg at a marked location on the vastus lateralis that would allow movement without interference from the NIRS device. A pulse oximeter (Caretaker, Caretaker Medical, USA) was used to measure SpO2 during HIIE. Blood lactate measurements (Lactate Plus, NOVA Biomedical, MA) were taken in duplicate at the ear lobe immediately before, and 5-minutes post HIIE.

Perceptual Measurement before and during HIIE Borg's rating of perceived exertion (6 rest to 20 maximal effort) scale (RPE) and thermal sensation (0 very cold to 8 very hot) was measured immediately before and every four minutes into HIIE. A breathlessness scale (0 mm no breathlessness to 200 mm maximal breathlessness)was used immediately before, at 10-minutes, and immediately after exercise to record subjective change in difficulty breathing. The highest measurements for both RPE (peak RPE) and thermal sensation (peak thermal sensation) were recorded per HIIE session performed. Additionally, RPE (RPE avg) and dyspnea scores were averaged over time for every HIIE session.

Thermal strain and hydration measurements During each HIIE exercise session continuous core temperature measurements were taken using rectal thermistors (Level 1 esophageal/rectal temperature probe, Smiths Medical, Minneapolis, MN, USA) connected to a thermometer (Precision 4000, YSI Incorporated, Yellow Springs, OH, USA) and monitored to ensure participant safety. Additionally, ∆ core temperature (i.e., the difference between peak core temperature and core temperature prior to starting exercise) and peak core temperature were recorded for each HIIE session. Sweat rate and dehydration were calculated from pre-exercise nude weight, post-exercise nude weight, water ingestion, and post-exercise urine output measurements27. Participants were asked to measure and report their pre-exercise and post-exercise nude weight using a digital scale (Cardinal DETECTO 758C, Webb City, MO) in a private room.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older and, are able to both speak and read in English.
* Physically active and used to high-intensity exercise.
* No known serious medical conditions.

Exclusion Criteria:

* Vulnerable populations such as children, minors, pregnant women, and intellectually challenged individuals.
* Those with cardiovascular, renal, metabolic, or chronic respiratory disease, smokers or those who have quit smoking less than 6 months ago, and those who use an inhaler to control for exercise-induced asthma.
* In addition, exclusion criteria include participants who show any signs or symptoms of COVID-19 and have had exposure to anyone with COVID-19 symptoms or any person that has tested positive for COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2021-06-11 (Actual); Study Completion 2021-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wells A, Fennel Z, Ducharme J, Masoud A, Houck J, Bellovary B, Deyhle M, Hsiao YY, Amorim F, Mermier C. Facemask Use During High Intensity Interval Exercise in Temperate and Hot Environments. J Occup Environ Med. 2022 May 1;64(5):421-428. doi: 10.1097/JOM.0000000000002461. Epub 2021 Dec 16. PMID 35608826

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded if in the last 6 months they smoked, performed less than 150 minutes of moderate-intensity exercise per week as defined by the American College of Sports Medicine guidelines, had a cardiorespiratory fitness classification below the 50th percentile for age and sex according to the American College Sport Medicine guidelines, reported no experience performing high intensity interval exercise, or had any known medical disease.
Groups:
- All Participants: Ten recreationally trained participants (5 males; 5 females) were recruited for this study. A randomized non-counterbalanced crossover repeated measures design was used to compare cardiovascular, thermoregulatory, metabolic, and perceived responses before and during high intensity interval exercise across four experimental trials performed during two visits with each visit lasting approximately 4 hours. For each high intensity interval exercise visit, which was separated by a minimum of 72 hours, the participants completed two high intensity interval exercise sessions separated by 3 hours of rest. The high intensity interval exercise sessions were performed in a temperate environment with and without a surgical mask, and in a hot environment with and without a surgical mask. During the 3-hour rest period participants were provided a 350-calorie meal (7 grams of Fat; 64 grams Carbohydrate; 9 grams of Protein) and water ad libitum.
Period: Overall Study
Arm/Group | All Participants
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participation in Four Different Conditions: Ten recreationally trained participants (5 males; 5 females) were recruited for this study. Participants were free from known cardiovascular, renal, metabolic, or chronic respiratory disease (i.e., asthma) as determined from a health history questionnaire. Participants were excluded if in the last 6 months they smoked and performed less than 150 minutes of moderate-intensity exercise per week, had a maximal oxygen consumption capacity below the 50th percentile for age and sex according to the American College of Sport Medicine guidelines for aerobic fitness, or reported no experience performing high intensity interval exercise. A pregnancy test was completed for female participants to include only non-pregnant participants.
  A randomized non-counterbalanced crossover repeated measures design was used to compare cardiovascular, thermoregulatory, metabolic, and perceived responses before and during high intensity across four experimental trials performed during two visits. The high intensity interval exercise sessions were performed in a temperate environment (23°C, 25% relative humidity) with and without a surgical mask, and in a hot environment (36°C, 14% relative humidity) with and without a surgical mask.
Arm/Group | Participation in Four Different Conditions
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.8 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Height (cm) [Mean (Standard Deviation); unit: centimeters] | 173.1 (7.5)
Weight (kg) [Mean (Standard Deviation); unit: kilograms] | 68.6 (11.5)
Resting SBP (mmHg) [Mean (Standard Deviation); unit: millimeters mercury] | 113.0 (8.0)
Resting DBP (mmHg) [Mean (Standard Deviation); unit: millimeters mercury] | 75.4 (5.9)
Resting HR (bpm) [Mean (Standard Deviation); unit: beats per minute] | 64 (9)
VO2max (mlO2/kg/min) [Mean (Standard Deviation); unit: mlO2/kg/min] | 49.4 (7.4)
Max Power (Watts) [Mean (Standard Deviation); unit: Watts] | 284.0 (78.0)

OUTCOME MEASURES:

1. Primary Outcome: Average Heart Rate Over the Course of High-intensity Interval Exercise
Description: Heart rate measured in beats per minute using a cardiograph impedance device (PhysioFlow)
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
beats per minute | 144 (21) | 143 (20) | 148 (18) | 149 (18)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental conditions; p = 0.003, 2x2 repeated measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.933, 2x2 repeated measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.344, 2x2 repeated measures ANOVA — A Bonferroni post-hoc test was used if significant interaction effect was present and p-values were adjusted based on the number of comparisons. To determine if a post-hoc was needed statistical significance was set to p < 0.05; No Method of Estimation was used

2. Primary Outcome: Average Stroke Volume Over the Course of High-intensity Interval Exercise
Description: Stroke volume measured in milliliters using a cardiograph impedance device (PhysioFlow)
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: milliliters
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
milliliters | 109.9 (19.5) | 109.2 (15.3) | 104.5 (16) | 101.5 (36.4)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; A 2x2 repeated measures ANOVA was performed to investigate statistical differences for all variables across the four conditions. Both main and interaction effects were calculated along with effect size, reported as partial ⴄ2 as provided by the statistical software JASP (version 0.14.1.0); Test type: Equivalence — Main effect for environmental conditions; p = 0.117, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.832, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.879, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

3. Primary Outcome: Average Cardiac Output Over the Course of High-intensity Interval Exercise
Description: Cardiac output measured in liters per minute using a cardiograph impedance device (PhysioFlow)
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
L/min | 15.7 (2.5) | 15.8 (2.6) | 15.3 (2.4) | 16.5 (2.2)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.749, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.311, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.368, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

4. Primary Outcome: Peak Core Temperature
Description: The highest core body temperature measured in degrees Celsius during high-intensity interval exercise
Time Frame: The highest value recorded during a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
°C | 37.76 (0.28) | 37.64 (0.29) | 37.65 (0.24) | 37.71 (0.38)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.789, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.739, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.158, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

5. Primary Outcome: Change From Baseline (Rest) in Core Temperature to the End of Exercise
Description: The difference in core temperature from rest prior to exercise and at the end of exercise
Time Frame: Baseline (rest) prior to exercise and immediately after 20-minutes of exercise
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
°C | 0.77 (0.22) | 0.54 (0.26) | 0.56 (0.20) | 0.64 (0.17)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.394, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.157, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.015, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

6. Primary Outcome: Sweat Rate During Exercise
Description: Amount of fluid loss through sweat over the course of exercise reported in milliliters per hour. This was calculated by taking difference of pre- and post-exercise body weight in kilograms while accounting for fluid intake and urine volume.
Time Frame: Change from Baseline (rest) prior to exercise and after 20-minutes of exercise
Measure: Mean (Standard Deviation); unit: milliliters per hour
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
milliliters per hour | 2097 (1258) | 1921 (690) | 2262 (1199) | 1793 (1254)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.960, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.073, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.503, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

7. Primary Outcome: Dehydration After Exercise
Description: Percentage of body weight fluid loss represented as a percentage of change from baseline and after 20 minutes of exercise
Time Frame: Change from baseline at rest and after 20-minutes of exercise
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
percentage of change | -0.76 (0.32) | -0.77 (0.26) | -0.81 (0.25) | -0.67 (0.28)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.786, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.180, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.239, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

8. Primary Outcome: Lactate at 5-minutes Post Exercise
Description: Blood lactate measured in millimoles per liter. This measurement was taken at the earlobe using a sterile lancet to obtain a drop of blood for analysis.
Time Frame: 5-minutes post exercise
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
mmol/L | 4.3 (1.7) | 4.2 (2.0) | 4.9 (2.2) | 4.5 (1.9)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.134, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.621, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.553, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

9. Primary Outcome: Average Blood Oxygen Saturation Over the Course of High-intensity Interval Exercise
Description: A pulse oximeter was placed on a finger and used to measure the percentage of oxygen saturated blood.
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: percent SpO2
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
percent SpO2 | 93.5 (3.63) | 93.7 (1.5) | 93.8 (2.3) | 94.0 (1.4)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.461, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.877, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.919, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

10. Primary Outcome: Average Muscle Tissue Oxygenation During the High-intensity Portions of the Exercise Session
Description: A near-infra red spectroscopy device was placed over the vastus lateralis of the dominant leg. This device measured the percentage of oxygenated muscle tissue.
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: percent SmO2
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
percent SmO2 | 31.0 (17.8) | 31.4 (21.5) | 23.5 (18.8) | 34.7 (21.7)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.466, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.186, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.080, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

11. Primary Outcome: Average Muscle Tissue Oxygenation During the Active Rest Portions of the Exercise Session
Description: as for outcome 10
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: percent SmO2
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
percent SmO2 | 56.7 (10.4) | 58.8 (15.9) | 55.8 (12.7) | 62.0 (11.4)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.375, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.178, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.533, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

12. Primary Outcome: Average Change in Muscle Tissue Oxygenation Between the Active Rest and High Intensity Portions Over the Course of High-intensity Interval Exercise.
Description: This value was calculated by subtracting the average percentage of muscle tissue oxygenation during active rest portion of the exercise from the average percentage of muscle tissue oxygenation during the high-intensity portion of the exercise.
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: percent SmO2
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
percent SmO2 | 25.6 (10) | 27.5 (10.2) | 32.4 (12.4) | 27.4 (13.7)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.290, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.527, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.045, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

13. Primary Outcome: Average Perceived Dyspnea Score Over the Course of High-intensity Interval Exercise
Description: The participants were presented a vertical 200 millimeter long line with the top of the line labeled "No Difficulty" and the bottom of the line labeled "Most Difficult". The participants were then asked to indicated on this line how difficult it was to breath by pointing to a point along the line presented to them. Once the participant indicated along the line how difficult it was to breath the researcher then marked the spot on the line with a pen. To quantify the measurement, the distance, measured in millimeters, was taken from the "No Difficulty" end of the line (0 millimeters) to the indicated mark with the maximum difficulty recorded as 200 millimeters.
Time Frame: Measurements were taken prior to, 10 minutes into exercise, and immediately after exercise (at 20 minutes). These measurements were averaged to form a single value for the high-intensity interval exercise session.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
units on a scale | 14 (13) | 44 (17) | 18 (15) | 58 (22)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.018, 2x2x3 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p < 0.001, 2x2x3 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.035, 2x2x3 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

14. Primary Outcome: Peak Thermal Sensation Over the Course of High-intensity Interval Exercise
Description: Participants were asked to indicate on a visual scale from 0 (very cold) to 8 (very hot) their perceived thermal sensation. The highest recorded value was reported.
Time Frame: Baseline (rest) and every four minutes that was assessed up to 20 minutes into exercise. The highest value was recorded for each exercise session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 5.9 (0.9) | 5.9 (0.9) | 6.5 (0.4) | 6.6 (0.4)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p < 0.001, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.678, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect; p = 0.678, 2x2 Repeated Measures ANOVA

15. Primary Outcome: Average Thermal Sensation Over the Course of High-intensity Interval Exercise
Description: Participants were asked to indicate on a visual scale from 0 (very cold) to 8 (very hot) their perceived thermal sensation.
Time Frame: Baseline (rest) and every four minutes that was assessed up to 20 minutes into exercise. These values were averaged into one value for each exercise session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 5.3 (0.7) | 5.4 (0.7) | 6.5 (0.4) | 6.6 (0.4)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p < 0.001, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.487, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.790, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

16. Primary Outcome: Peak Rating of Perceived Exertion Over the Course of High-intensity Interval Exercise
Description: Participants were asked to indicate on a visual scale from 6 (no exertion) to 20 (maximal exertion) their perceived difficulty of exercise. The highest recorded value was reported.
Time Frame: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 15 (2) | 15 (1) | 15 (2) | 16 (2)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.089, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.297, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.111, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

17. Primary Outcome: Averaged Rating of Perceived Exertion Over the Course of High-intensity Interval Exercise
Description: as for outcome 16
Time Frame: Baseline (rest) and every four minutes that assessed up to 20 minutes into exercise. These values were averaged into one value for each exercise session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
score on a scale | 13.3 (1.4) | 13.3 (1.2) | 13.5 (1.2) | 14.3 (1.3)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.024, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.002, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.014, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

18. Primary Outcome: Peak Heart Rate Over the Course of High-intensity Interval Exercise
Description: Peak heart rate measured in beats per minute using a cardiograph impedance device (PhysioFlow)
Time Frame: During a 20-minute high-intensity interval exercise session
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
Number analyzed (Participants) | 10 | 10 | 10 | 10
beats per minute | 164 (20) | 164 (17) | 169 (16) | 169 (16)
Statistical Analysis 1: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for environmental condition; p = 0.012, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 2: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Main effect for mask condition; p = 0.893, 2x2 Repeated Measures ANOVA — Statistical significance was set at p < 0.05
Statistical Analysis 3: Comparison: No Mask Temperate vs Mask Temperate vs No Mask Hot vs Mask Hot; Test type: Equivalence — Interaction effect across environmental and mask conditions; p = 0.969, 2x2 Repeated Measures ANOVA — [p-value comment as in outcome 1, analysis 3]

ADVERSE EVENTS:
Time Frame: up to 4 weeks
Groups:
- No Mask Temperate: High-intensity interval exercise without using a surgical face mask in a temperate environment Participants performed high-intensity interval exercise in a temperate environmental condition without wearing a surgical face mask.
- Mask Temperate: Device: High-intensity interval exercise with surgical face mask in a temperate environment Participants performed high-intensity interval exercise in a temperate environmental condition while wearing surgical face mask
- No Mask Hot: High-intensity interval exercise without using a surgical face mask in a hot environment Participants performed high-intensity interval exercise in a hot environmental condition without wearing a surgical face mask.
- Mask Hot: Device: High-intensity interval exercise with surgical face mask in a hot environment Participants performed high-intensity interval exercise in a hot environmental condition while wearing surgical face mask
Arm/Group | No Mask Temperate | Mask Temperate | No Mask Hot | Mask Hot
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
The current study design employed a three-hour rest between same day trials. Thus, the fatigue from the first trial may have carried over to the second trial. However, this limitation was thought to be minimized as the trial order was randomized, the participants were aerobically fit individuals, and only a total of 5 minutes was spent exercising at 85% of their maximum power output per trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT05143801/Prot_SAP_002.pdf
  • Informed Consent Form (2022-02-26): https://cdn.clinicaltrials.gov/large-docs/01/NCT05143801/ICF_003.pdf